CLINICAL TRIAL: NCT01799902
Title: Belgian Observational Study to Evaluate Storage and Voiding Symptoms Improvement in Male Subjects With Lower Urinary Tract Predominant Storage Symptoms (Overactive Bladder Syndrome) Being Treated With Solifenacin in Monotherapy or Combination
Brief Title: Treatment of Symptoms in Male Patients With Lower Urinary Tract Symptoms (LUTS) Predominant Storage Symptoms (Overactive Bladder Syndrome)
Acronym: VENICE
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Veeda Clinical Research (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: BE-11-VES-01
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Lower Urinary Tract Predominant Storage Symptoms
Keywords: Observational; Non-Interventional Prospective; Phase IV Treatment; Overactive Bladder Syndrome; Solifenacin
MeSH Terms: interventions — Solifenacin Succinate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Male subjects with LUT predominant storage symptoms (OAB): male subjects with Overactive Bladder Syndrome (OAB) being treated with solifenacin in monotherapy or combination
  Interventions: Drug: Solifenacin

INTERVENTIONS:
Drug: Solifenacin — Oral
  Other Names: YM905, Vesicare®

SUMMARY:
This study is a non interventional study where no investigational medicine is provided. Procedures and examination will follow the institution standard of care practice. The therapeutic approach will not be decided in advance by the protocol or influenced in any way by the protocol.

After standard evaluation the investigator will decide the treatment strategy and upon eligibility criteria met will propose subject to participate to the study. Informed consent will be collected for all subjects.

The study will consist of 3 possible observational visits; V1 (enrolment), V2 and V3 (follow up).

During all observational visits (V1, V2 and V3) the patient will complete the I-PSS (International Prostate Symptom Score) questionnaire including Quality Of Life (QOL) questionnaire and a Patient assessment of treatment benefit and satisfaction using a Visual Analogue Scale (VAS).

The patient will be asked to complete a voiding diary the first 3 days after Visit 1 (Baseline diary), 3 days before Visit 2 and again 3 days before Visit 3.

Prostate Specific Antigen (PSA) measurement- Uroflowmetry - Post Voiding Residual volume and Trans Rectal Ultra Sound data will be collected only if available.

During all observational visits (V1, V2 and V3) the investigator will complete the assessment of treatment benefit and satisfaction using a VAS.

ELIGIBILITY:
Inclusion Criteria:

The following subjects can be included in this study if they answer the following criteria:

* they have been prescribed solifenacin 5-10mg according to Summary of Product Characteristics (SmPC).
* Subjects with diagnosed Lower Urinary Tract Symptoms (LUTS) with substantial storage disorder defined as urgency, and/or frequency and/or Urge Urinary Incontinence (UUI) at the discretion of the investigator.
* IPSS storage sub-score > 8
* Subject expected to require at least 3 months treatment with solifenacin.

Exclusion Criteria:

* Any reason which following current medical knowledge, physical condition of the patient and in the opinion of the investigator contraindicates administration of solifenacin to the subject, such as- signs and symptoms suggestive of urinary tract infection (confirmed by positive urine analysis).
* History of bladder obstruction not being adequately corrected.
* Anticipate or plan to participate in another study during study period of 12 weeks from study entry.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients in Belgium with lower urinary tract predominant storage symptoms (Overactive Bladder Syndrome) being treated with solifenacin in monotherapy or combination.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2011-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in I-PSS storage scores (frequency, urgency, nocturia) | Baseline, Week 6 and 12
  To evaluate the effect of solifenacin monotherapy or combination with an α receptor blocker on storage symptoms measured by the patient I-PSS (International Prostate Symptom Score questionnaire)

SECONDARY OUTCOMES:
Change in Storage symptoms assessed in the patient bladder diary by Mean number of micturitions per 24 hours | Baseline, Week 6 and 12
Change in Storage symptoms assessed in the patient bladder diary by Mean number of incontinence episodes per 24 hours | Baseline, Week 6 and 12
Change in Storage symptoms assessed in the patient bladder diary by Mean number of urgency (grade 3 or 4, Patient Perception of Intensity of Urgency Scale (PPIUS)) episodes per 24 hours | Baseline, Week 6 and 12
Change in Storage symptoms assessed in the patient bladder diary by Mean number of urge incontinence (grade 4, PPIUS) episodes per 24 hours | Baseline, Week 6 and 12
Voiding scores (incomplete emptying, intermittency, weak stream and straining) | Week 1, 6 and 12
Total and individual I-PSS item scores | Week 1, 6 and 12
Quality Of Life assessed by the patient I-PSS questionnaire | Week 1, 6 and 12
Treatment satisfaction and treatment benefit for investigator using a visual analogue scale (VAS) | Week 1, 6 and 12
Treatment satisfaction and treatment benefit for patient using a visual analogue scale (VAS) | Week 1, 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe B.V.
Locations (15):
- Belgium (15):
  - ASZ, Aalst
  - ZNA Stuyvenberg, Antwerp
  - Erasme, Brussels
  - UZ Brussel, Brussels
  - Private practice, Brussels
  - AZ St. Monica, Deurne
  - UZ Antwerpen, Edegem
  - Maria Middelares, Ghent
  - Sint-Lucas, Ghent
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - AZ Damiaan, Ostend
  - AZ Oudenaarde, Oudenaarde
  - H.Hart Roeselaere, Roeselaere
  - AZ Sint Elisabeth, Zottegem